CLINICAL TRIAL: NCT02597803
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of RGN-259 Ophthalmic Solutions for the Treatment of Dry Eye: ARISE-1
Brief Title: Assessment of the Safety and Efficacy of RGN-259 Ophthalmic Solutions for Dry Eye Syndrome: ARISE-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ReGenTree, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-259
Record Dates: First submitted 2015-10-26; First posted 2015-11-05 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Dry Eye; DES
MeSH Terms: conditions — Dry Eye Syndromes | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose RGN-259 (Experimental): High dose RGN-259: It is a preservative-free, sterile eye drop solution containing Tβ4
  Interventions: Drug: RGN-259
- Placebo (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Interventions: Drug: Placebo
- Low Dose RGN-259 (Experimental): Low dose RGN-259: It is a preservative-free, sterile eye drop solution containing Tβ4
  Interventions: Drug: RGN-259

INTERVENTIONS:
Drug: RGN-259 — A preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into each eye, four times a day (QID) for 28 days
  Other Names: Tβ4; Thymosin Beta 4
  Arms: High Dose RGN-259; Low Dose RGN-259
Drug: Placebo — It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of RGN-259 Ophthalmic Solutions to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
Dry eye can be caused by many variable factors. Some examples include hormonal changes due to aging, or living in an environment of low humidity for long periods of time. Dry eye is a complex disease that may result in symptoms like discomfort, visual disturbance, and dryness. Patients with dry eye often have damage on the surface of the eye. In previous studies, RGN-259 has been shown to promote healing of the surface of the eye and decrease inflammation. It suggests that RGN-259 has a significant potential to be an important new safe and effective therapeutic in the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye for at least 6 months
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months
* Have a Schirmer's Test score of ≤10mm and ≥1mm
* Have a Tear Film Break-Up Time (TFBUT) ≤10 seconds
* Have a corneal fluorescein staining score of ≥2 in at least one region of the cornea

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 6 months;
* Have an IOP > 25 mmHg at Visit 1;
* Have any planned ocular and/or lid surgeries over the study period;
* Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;
* Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study);
* Have corrected visual acuity greater than or equal to logMAR +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total corneal fluorescein staining score at day29 | 29 days after first dosing
Total ocular discomfort score at day29 | 29 days after first dosing

SECONDARY OUTCOMES:
Tear film break-up time at day 8, 15, 29 | 8, 15, 29 days after first dosing
Unanesthetized Schirmer's Test at day 8, 15, 29 | 8, 15, 29 days after first dosing
Ocular Surface Disease Index (OSDI)© at day 8, 15, 29 | 8, 15, 29 days after first dosing

OTHER OUTCOMES:
Visual acuity ( ETDRS, Early Treatment Diabetic Retinopathy Study scale) at 1, 8, 15, 29 days after first dosing | 1, 8, 15, 29 days after first dosing
Change in biomicroscopy using slit-lamp at 8, 15, 29 days after first dosing | 1, 8, 15, 29 days after first dosing
Corneal Sensitivity (aesthesiometer (Cochet-Bonnet at 1, 8, 15, 29 days after first dosing | 1, 8, 15, 29 days after first dosing
Adverse event query at Visits 1,2,3, 4 and 5 | 1, 8, 15, 29 days after first dosing
Change in biomicroscopy using Undilated Fundoscopy at 1, 29 days after first dosing | 1, 29 days after first dosing
Intraocular Pressure at Visits 1, 29 days after first dosing | 1, 29 days after first dosing

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Ora Clinical Research and Development
Locations (1):
- Andover, MA, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No